CLINICAL TRIAL: NCT01872806
Title: Radiation Meter Controlled Electrophysiological Reactivity (EEG and ECG) Due to Mobile Phone Radiation.
Brief Title: Electrophysiological Reactivity Due to Mobile Phone Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: METC azM/UM NL44004.068.13
Record Dates: First submitted 2013-05-30; First posted 2013-06-07 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Mobile phone radiation (Experimental): Dialing mobile phone placed against the ear/chest for a duration of 15 minutes, before and after 15 minutes sham phone will be placed against the ear/chest.
  Interventions: Radiation: a dialing smartphone will be placed on the chest and the ear

INTERVENTIONS:
Radiation: a dialing smartphone will be placed on the chest and the ear

SUMMARY:
The main objective of this study is to investigate whether radiofrequency electromagnetic radiation, induced by a dialing mobile phone placed on the body, causes a change in electrophysiology.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether placement of a 3G dialing mobile phone causes direct changes in EEG activity compared to the placement of a sham phone. Furthermore, it is investigated whether placement of the mobile phone on the ear or the heart results in different outcomes. The subjects are measured twice: on one of the two days the mobile phone is attached to the ear, the other day to the chest. In this single-blind, cross-over design, assessments in the sham phone conditions are conducted directly preceding and following the mobile phone exposure. During each assessment, EEG activity and radiofrequency radiation are recorded jointly. Delta, theta, alpha, slowbeta, fastbeta, and gamma activity are computed. The association between radiation exposure and the EEG is tested using multilevel random regression analyses with radiation as predictor of main interest.

ELIGIBILITY:
Inclusion Criteria:

* female aged between 18 - 30 years

Exclusion Criteria:

* cardiac or brain disorder
* pregnancy

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in EEG and ECG | during mobile phone exposure (immediately)

CONTACTS AND LOCATIONS:
Overall Officials: Jim van Os, Principal Investigator — Maastricht University
Locations (1):
- Mondriaan, locatie Vijverdal, Maastricht University, Maastricht, Limburg, Netherlands